CLINICAL TRIAL: NCT05625633
Title: Human Papillomavirus (HPV) Vaccination for the Treatment of Refractory Cutaneous Warts: A Randomized, Placebo-Controlled, Double-Blinded Trial
Brief Title: Human Papillomavirus (HPV) Vaccination vs. Placebo for the Treatment of Refractory Cutaneous Warts
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Western Institute for Veterans Research (Other)
Collaborators: University of Utah (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00152954
Record Dates: First submitted 2022-11-07; First posted 2022-11-23 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Warts
Keywords: Refractory cutaneous warts; Human Papillomavirus (HPV) Vaccination; HPV vaccine
MeSH Terms: conditions — Warts; Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine nonavalent; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and Nurses share the role as Care Provider. Investigators will be blinded to the treatment allocation. Nurses, however, will be aware of the treatment allocation as they are administering the injections. Nurses are not involved in the study conduct in any other way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HPV Vaccine (Experimental): 0.5-mL suspension of 9-valent Gardasil vaccine administered as intramuscular injection at weeks 0, 4, and 20
  Interventions: Biological: Human Papillomavirus 9-valent Vaccine, Recombinant
- Placebo (Placebo Comparator): 0.5-mL normal saline administered as intramuscular injection at weeks 0, 4, and 20
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Human Papillomavirus 9-valent Vaccine, Recombinant — 0.5-mL suspension of 9-valent Gardasil administered as intramuscular injection at weeks 0, 4, and 20
  Other Names: Gardasil 9; 9-valent Gardasil
  Arms: HPV Vaccine
Other: Normal Saline — 0.5-mL normal saline administered as intramuscular injection at weeks 0, 4, and 20
  Arms: Placebo

SUMMARY:
This double-blinded clinical trial randomly assigns participants with refractory cutaneous warts to receive either treatment with the human papillomavirus (HPV) vaccine or a placebo to assess the efficacy of HPV vaccination for the treatment of refractory cutaneous warts.

DETAILED DESCRIPTION:
Cutaneous warts are a common cause for medical office visits and are frequently encountered in dermatology practice. Despite their benign nature, cutaneous warts can be painful, disfiguring, persistent and may be associated with significant morbidity. Numerous therapeutic options are available, including local destruction, virucidal agents, topical and systemic antiproliferative medications, and immunotherapy. Unfortunately, no single therapy is uniformly effective, and patients often receive multiple courses of treatment (cryotherapy, curettage, Candida antigen injection, etc.) without improvement.

An efficacious therapy for cutaneous warts is sorely needed and treatment with HPV vaccination is being increasingly reported. Notably, individual cases and case series have reported complete resolution of multiple treatment refractory warts after treatment with the quadrivalent HPV vaccine. Even more encouraging, a larger retrospective study of 30 patients found that up to 60% of patients had a complete or partial response after treatment with the HPV vaccine. Additional benefits of treatment with HPV vaccination include ease of use, less tissue destruction and pain, and the potential for less frequent medical office visits. Despite these promising preliminary data, a larger, randomized controlled study has yet to be performed.

This will be a multi-center, double-blinded, randomized, placebo-controlled trial with 120 participants. Enrolled participants will be randomized to treatment with either HPV vaccination or placebo. Participants will receive injections with the 9-valent HPV vaccine or placebo at 0, 4, and 20 weeks and follow up until 24 weeks to determine their treatment response, quality of life and the safety and tolerability of HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and provide written informed consent
2. Age 18 or older
3. Clinical diagnosis of cutaneous warts
4. Must have received prior treatment for cutaneous warts (such as curettage, cryotherapy, salicylic acid, intralesional Candida antigen injection, etc.)

Exclusion Criteria:

1. Untreated cutaneous warts
2. Anogenital warts
3. Oral warts
4. Treatment for cutaneous warts in the past 4 weeks
5. Active acute illness
6. Immunosuppression
7. Known hypersensitivity to HPV vaccination
8. Subjects may not receive any other investigational treatment
9. Pregnancy or planned pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessing the efficacy/therapeutic response of HPV vaccination for the treatment of refractory cutaneous warts (response information may be found in description) at 24 weeks | Response to treatment assessments will occur 24 weeks after first dose of vaccine/placebo (primary endpoint)
  Assessing the efficacy/therapeutic response of HPV vaccination for the treatment of refractory cutaneous warts, classified as: (1) complete response (CR; complete clearance of warts); (2) partial response (PR; any decrease in lesion number or size); or (3) no response (NR; no change or increase in lesion number or size)
Assessing the efficacy/therapeutic response of HPV vaccination for the treatment of refractory cutaneous warts (response information may be found in description) at 4 weeks | Response to treatment assessments will occur 4 weeks after first dose of vaccine/placebo
  Assessing the efficacy/therapeutic response of HPV vaccination for the treatment of refractory cutaneous warts, classified as: (1) complete response (CR; complete clearance of warts); (2) partial response (PR; any decrease in lesion number or size); or (3) no response (NR; no change or increase in lesion number or size)
Assessing the efficacy/therapeutic response of HPV vaccination for the treatment of refractory cutaneous warts (response information may be found in description) at 8 weeks | Response to treatment assessments will occur at 8 weeks after first dose of vaccine/placebo
  Assessing the efficacy/therapeutic response of HPV vaccination for the treatment of refractory cutaneous warts, classified as: (1) complete response (CR; complete clearance of warts); (2) partial response (PR; any decrease in lesion number or size); or (3) no response (NR; no change or increase in lesion number or size)

SECONDARY OUTCOMES:
Skindex-16 | Quality of life assessments will occur at 0 (baseline), 4, 8, and 24 weeks (primary endpoint)
  Assessing for changes in quality of life, as indicated by the Skindex-16 questionnaire
Incidence of Treatment-Emergent Adverse Events | Safety assessment will occur at 0, 4, 8, 20, and 24 weeks
  Assessing the safety and tolerability of HPV vaccination via adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Lowell Nicholson, MD, Principal Investigator — University of Utah Health Care System
Locations (2):
- United States (2):
  - University of Utah Midvalley Health Center, Salt Lake City, Utah
  - VA Salt Lake City Health Care System, Salt Lake City, Utah